CLINICAL TRIAL: NCT00624637
Title: Does Massage With or Without Aromatherapy Reduce Infant's Distress After Craniofacial Surgery? A Randomized Controlled Trial
Brief Title: Does Massage With or Without Aromatherapy Reduce Infant's Distress?
Acronym: aromatherapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Dr Monique van Dijk, Erasmus MC-Sophia Children's Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2007-253
Record Dates: First submitted 2008-02-15; First posted 2008-02-27 (Estimated); Last update posted 2008-02-27 (Estimated); Status verified 2008-02

CONDITIONS: Distress
Keywords: aromatherapy; massage; comfort; postoperative; infants; craniofacial surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Other): infants after craniofacial surgery receive one massage with aromatherapy three hours postoperatively
  Interventions: Other: aromatherapy massage
- B (Other): infants after craniofacial surgery receive one massage with carrier oil three hours postoperatively
  Interventions: Other: aromatherapy massage
- C (No Intervention): no intervention, standard postoperative care

INTERVENTIONS:
Other: aromatherapy massage — Ten minutes massage of hands, arms or feet with mandarin essential oil 1% (Citrus reticulata) or with carrier oil only
  Other Names: A - aromatherapy massage; B - massage
  Arms: A; B

SUMMARY:
This study aims to determine the effect of massage with or without aromatherapy on infant´s level of distress

DETAILED DESCRIPTION:
Despite extensive use of pharmacological treatments such as sedatives, distress and anxiety remain a huge problem in patients admitted to the PICU, especially in the 65% under the age of 3. Parents are anxious about the outcome and feel powerless because they have to transfer care to doctors and nurses. Those in favor of complementary care, realize at the same time that there is lack of evidence to support its use in daily practice. On the other hand, many sedatives used in infants are unlicensed and animal studies even suggest increased risk of neuroapoptosis using midazolam at an early age.

In a first study we will evaluate the effects of aromatherapy massage or massage compared to standard care in infants after craniofacial surgery.

The first group receives: aromatherapy massage using a concentration of mandarin essence in the massage oil, the second group: massage (without essential oils) and the third (control) group receives standard postoperative care. Massage will be performed in a standardized way using the ' m' technique® developed by dr. Buckle. Primary outcome is the percentage of patients with COMFORT behavior score below 17, assessed from videomaterial by a rater blinded for condition.The intervention will be carried out three hours after return from surgery.Secondary outcomes are bedside COMFORT behavior scores assessed by the caregiving nurse and the amount of midazolam used in the first 24 hours postoperative as well as the use of additional analgesics such as paracetamol and morphine.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged 6 to 36 months admitted to the Intensive Care-Sophia after craniofacial surgery

Exclusion Criteria:

* Neurological impairment
* Eczema or other skin disorders
* Nut allergy

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
level of COMFORT with videotaped COMFORT behavior scale | first 24 hours postoperative

SECONDARY OUTCOMES:
COMFORT behavior bedside and Visual Analogue Scale distress, change in Heart Rate, change in Mean Arterial Pressure, amount of required sedatives/opioids | first 24 hours postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Dick Tibboel, prof, MD, Study Director — Erasmus MC-Sophia
Locations (1):
- Pediatric Surgical Intensive Care, Erasmus MC-Sophia, Rotterdam, South Holland, Netherlands

REFERENCES:
- [Derived] de Jong M, Lucas C, Bredero H, van Adrichem L, Tibboel D, van Dijk M. Does postoperative 'M' technique massage with or without mandarin oil reduce infants' distress after major craniofacial surgery? J Adv Nurs. 2012 Aug;68(8):1748-57. doi: 10.1111/j.1365-2648.2011.05861.x. Epub 2011 Nov 3. PMID 22050553